CLINICAL TRIAL: NCT05246358
Title: Respiratory Rate Validation Study - ChroniSense Polso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChroniSense Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR 2020-414
Record Dates: First submitted 2022-01-23; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ChroniSense Polso Respiratory Rate (Experimental): Comparison of respiratory rates in normal subjects as observational with end tidal CO2. No treatment or interventions will be performed
  Interventions: Device: ChoniSense Polso

INTERVENTIONS:
Device: ChoniSense Polso — A range of stable respiratory rates was elicited from each volunteer test subject. The rates were 5, 10, 15, 20, 25, 30, 35, 40 and 45 breaths per minute; with some natural variation from these exact numbers.
  Each subject was instrumented with an open system mask that allows for measurement of the end tidal carbon dioxide (EtCO2) respiratory rate and tidal volume. The EtCO2 monitor was used as the Accuracy Reference Device (Reference) in this study.

SUMMARY:
20 volunteer test subjects entered into an accuracy study that is designed to validate accuracy of the respiratory rate of the ChroniSense Polso

DETAILED DESCRIPTION:
20 volunteer test subjects entered into an accuracy study that is designed to validate accuracy of the respiratory rate of the ChroniSense Polso.

A range of stable respiratory rates were elicited from each volunteer test subject. The rates will be approximately 5, 10, 15, 20, 25, 30, 35, 40 and 45 breaths per minute; with some natural variation from these exact numbers.

Each subject was instrumented with an open system mask that allows for measurement of the end tidal carbon dioxide (EtCO2) respiratory rate and tidal volume. The EtCO2 monitor was used as the Accuracy Reference Device (Reference) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is adult over 18 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker, or a smoker who has refrained from smoking for 1 day.
* Male or female of any race

Exclusion Criteria:

Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoo in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)

* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with self-reported heart or cardiovascular conditions such as:

  * high blood pressure: systolic >140 mmHg or diastolic >90 mmHg
  * have had cardiovascular surgery
  * chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease, kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
  * Cancer / chemotherapy
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Arms accuracy (breaths per minute) of Polso Monitoring System relative to End Tidal Carbon Dioxide monitor-derived respiration rate | Through study completion, 1 month average
  Accuracy of Polso Monitoring System (DUT) relative to a reference End Tidal Carbon Dioxide monitor-derived respiration rate (REF). Polso reports respiration rate (breaths per minute) directly, at 60 second intervals. End Tidal Carbon Dioxide monitor waveforms will be hand-scored, based on respiration waveform peaks, to derive respiration rate (breaths per minute). The readings from each device will be synchronized to achieve paired simultaneous respiration rates, and aggregated into calculation of a comparative accuracy measure, namely Accuracy root-mean-square (Arms) difference, in breaths per minute, between the Polso (DUT) and the reference (REF) respiratory rate system, for all stable respiratory periods. Acceptance criteria Arms <3.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark Desaturation Laboratory, Site ID# 001, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No